CLINICAL TRIAL: NCT00524615
Title: Addition of Spironolactone in Patients With Resistant Arterial Hypertension
Acronym: ASPIRANT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jan Vaclavík (Other)
Collaborators: Czech Society of Hypertension (Other); Prostejov Hospital (Unknown); Brno University Hospital (Other); Olomouc Military Hospital (Unknown); Gedeon Richter Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Jan Vaclavík, Principal investigator, University Hospital Olomouc
Organization: University Hospital Olomouc (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASPIRANT-1; EudraCT 2007-003558-27
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Hypertension
Keywords: resistant hypertension treatment; spironolactone; aldosterone antagonists; resistant arterial hypertension; refractory arterial hypertension
MeSH Terms: conditions — Hypertension | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 25 mg of Spironolactone oraly once daily
  Interventions: Drug: spironolactone
- 2 (Placebo Comparator): placebo oraly once daily
  Interventions: Drug: spironolactone

INTERVENTIONS:
Drug: spironolactone — 25 mg of spironolactone once daily or placebo for 2 months

SUMMARY:
The purpose of this study is to evaluate the efficacy of spironolactone on lowering blood pressure when added to therapy in patients with resistant arterial hypertension.

DETAILED DESCRIPTION:
Arterial hypertension resistant to therapy and requiring treatment with more then three antihypertensive drugs is common. At present there are is no standard therapy for resistant hypertension based on randomised clinical trials, neither data to guide addition of further drugs to therapy. Recently some observational and retrospective trials reported good effect of spironolactone in patients with resistant hypertension, but these data were not validated by prospective randomised clinical trials.

This is a multicentric, randomised, double blind clinical trial, which will evaluate the effect of addition of 25 mg spironolactone to current medication compared to placebo. The study will enroll patients with blood pressure over 140/90 mmHg during a clinical examination, which are using at least three antihypertensive drugs, one of them being a diuretic. Average daytime systolic and diastolic blodd pressure will be evaluated by ABPM (ambulatory blood pressure monitoring).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Resistant arterial hypertension: (blood pressure during clinical control exceeding 140/90 mmHg (or 130/80 mmHg in in diabetic patients or patients with renal disease with creatinine level of more than 133 μmol per liter or urinary protein excretion of more than 300 mg over a 24-hour period) despite adherence to treatment with full doses of at least three antihypertensive medications, including a diuretic

Exclusion Criteria:

* Pregnant or breastfeeding women, women in fertile age without ruled out pregnancy
* Severe hypertension over 180/110 mmHg
* Renal insufficiency with creatinine over 180 umol/l or GFR lower than 40 ml/min
* Hyperkalemia over 5,4 mmol/l, hyponatremia below 130 mmol/l
* Porphyria
* Hypersensitivity to the compounds of Verospiron (Richter Gedeon, Hungary) drug
* Patients taking any aldosterone antagonist (spironolactone, eplerenone, kanreone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2007-09; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Average daytime systolic and diastolic blodd pressure evaluated by ABPM (ambulatory blood pressure monitoring) | before and after 2 months of treatment

SECONDARY OUTCOMES:
changes of serum potassium, natrium, creatinine, body weight, casual blood pressure in office, treatment response for different baseline levels of aldosterone and aldosterone/PRA ratio | 2 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jan Václavík, MD., Study Director — Internal medicine department I, Olomouc university hospital and Palacký University School of medicine; Bořek Lačňák, MD., Principal Investigator — Internal Medicine Dept., Šternberk Hospital; Martin Plachý, MD., Principal Investigator — Internal medicine department II, Brno University Hospital
Locations (1):
- Olomouc University Hospital and Palacký University School of Medicine, Olomouc, Czechia

REFERENCES:
- [Background] Chapman N, Dobson J, Wilson S, Dahlof B, Sever PS, Wedel H, Poulter NR; Anglo-Scandinavian Cardiac Outcomes Trial Investigators. Effect of spironolactone on blood pressure in subjects with resistant hypertension. Hypertension. 2007 Apr;49(4):839-45. doi: 10.1161/01.HYP.0000259805.18468.8c. Epub 2007 Feb 19. PMID 17309946
- [Background] Sharabi Y, Adler E, Shamis A, Nussinovitch N, Markovitz A, Grossman E. Efficacy of add-on aldosterone receptor blocker in uncontrolled hypertension. Am J Hypertens. 2006 Jul;19(7):750-5. doi: 10.1016/j.amjhyper.2005.11.016. PMID 16814132
- [Derived] Vaclavik J, Sedlak R, Jarkovsky J, Kocianova E, Taborsky M. Effect of spironolactone in resistant arterial hypertension: a randomized, double-blind, placebo-controlled trial (ASPIRANT-EXT). Medicine (Baltimore). 2014 Dec;93(27):e162. doi: 10.1097/MD.0000000000000162. PMID 25501057
- [Derived] Vaclavik J, Sedlak R, Plachy M, Navratil K, Plasek J, Husar R, Kocianova E, Taborsky M. Addition of spironolactone in patients with resistant arterial hypertension (ASPIRANT)--study protocol. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2011 Jun;155(2):143-8. doi: 10.5507/bp.155.2011.004. PMID 21804623
- [Derived] Vaclavik J, Sedlak R, Plachy M, Navratil K, Plasek J, Jarkovsky J, Vaclavik T, Husar R, Kocianova E, Taborsky M. Addition of spironolactone in patients with resistant arterial hypertension (ASPIRANT): a randomized, double-blind, placebo-controlled trial. Hypertension. 2011 Jun;57(6):1069-75. doi: 10.1161/HYPERTENSIONAHA.111.169961. Epub 2011 May 2. PMID 21536989
- See also: Palacký University School of Medicine — http://www.lf.upol.cz/en/
- See also: Olomouc University Hospital — http://www.fnol.cz/